CLINICAL TRIAL: NCT06004414
Title: Hybrid Type I Effectiveness-implementation Trial of SilverCloud as a School-based Intervention for Vulnerable Youth
Brief Title: SilverCloud as a School-Based Intervention for Vulnerable Youth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-00257
Record Dates: First submitted 2023-08-17; First posted 2023-08-22 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Depression; Anxiety
Keywords: depression; anxiety; behavioral therapy
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- SilverCloud (Experimental): Adolescents who seek or are referred for mental health services and screen positive for significant mental health symptoms randomized to receive SilverCloud.
  Interventions: Behavioral: App-based Cognitive Behavioral Therapy (CBT)
- Treatment as Usual (TAU) (Active Comparator): Adolescents who seek or are referred for mental health services and screen positive for significant mental health symptoms randomized to receive psychotherapy.
  Interventions: Behavioral: Psychotherapy

INTERVENTIONS:
Behavioral: App-based Cognitive Behavioral Therapy (CBT) — SilverCloud is organized into eight core modules that follow evidence-based principles of CBT, along with six additional modules that can be prescribed by the clinician to address a participant's specific needs.
  Other Names: SilverCloud
  Arms: SilverCloud
Behavioral: Psychotherapy — Psychotherapy with a licensed clinician at one of the study sites.
  Arms: Treatment as Usual (TAU)

SUMMARY:
The goal of this study is to test the efficacy and feasibility of a clinician-guided, app-based cognitive behavioral therapy (CBT) program, SilverCloud, as a school-based mental health intervention for vulnerable youth. An open trial of SilverCloud will be conducted to determine preliminary efficacy in this sample and inform program refinements by collecting outcome self-report assessments and conducting interviews on feasibility and acceptability. After the program and its implementation strategy are refined, we will conduct an randomized controlled trial. Adolescents who seek or are referred for mental health services through one of the study sites and screen positive for significant mental health symptoms will be randomized to receive SilverCloud or treatment as usual (TAU). Efficacy will be assessed through outcome self-reports. Feasibility and acceptability feedback will again be collected from participants, SBHC staff, and community members.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in the phase I open trial of this study, an individual must meet all of the following criteria:

* Enrolled in a high school
* Score of 10+ on GAD-7 or PHQ-9
* Speak/read English. The current investigational version of SilverCloud that will be used in this study is only available in English.

In order to be eligible to participate in the RCT of this study, an individual must meet all of the following criteria:

* Enrolled in 9th through 11th grades.
* Score of 10+ on GAD-7 or PHQ-9
* Enrolled in one of the study sites
* Speak/read English. The current investigational version of SilverCloud that will be used in this study is only available in English.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in the phase I open trial of this study:

* Does not use a smartphone
* Mental health concerns for which intensive treatment is indicated. Because SilverCloud has not been evaluated in people with serious mental illness, participants who exhibit symptoms of mania or psychosis will be referred to a higher level of care.
* Current suicidal ideation with intent. Participants who have a suicide plan and intent to act on it will be referred to the SBHC suicide risk protocol and will not be eligible until their suicidal thoughts have abated.

An individual who meets any of the following criteria will be excluded from participation in the RCT of this study:

* Current (within 1 month of enrollment) mental health treatment at one of the study sites
* Does not use a smartphone
* Mental health concerns for which intensive treatment is indicated. Because SilverCloud has not been evaluated in people with serious mental illness, participants who exhibit symptoms of mania or psychosis will be referred to a higher level of care.
* Current suicidal ideation with intent. Participants who have a suicide plan and intent to act on it will be referred for crisis intervention through the site at which they were referred and will not be eligible until their suicidal thoughts have abated.

Ages: 13 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 (PHQ-9) Score | Baseline, Week 8
  The PHQ-9 is a 9-item questionnaire assessing the degree of depression severity. Items are ranked on a 4-point scale ranging from 0 (not at all) to 3 (nearly every day). The total score is the sum of responses and ranges from 0-27; higher scores indicate greater severity of depression.
Change in General Anxiety Disorder-7 (GAD-7) Score | Baseline, Week 8
  The GAD-7 is a 7-item questionnaire assessing the degree of anxiety severity. Items are ranked on a 4-point scale ranging from 0 (not at all) to 3 (nearly every day). The total score is the sum of responses and ranges from 0-21; higher scores indicate greater severity of anxiety.

SECONDARY OUTCOMES:
Change in Revised Children's Anxiety and Depression Scale (RCADS-25) Youth Self-Report Score | Baseline, Week 8
  The RCADS-25 is a self-report questionnaire that assesses symptoms of depression and anxiety in children and adolescents. Each item is rated as 0 (never), 1 (sometimes), 2 (often), or 3 (always). The raw score is the sum of responses and is converted to a T-score where: below 65 = normal range; between 65-69 = borderline clinical range; and 70 above = clinical range.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Item Bank v2.0 - Peer Relationships - Short Form 8a Score | Baseline, Week 8
  This is an 8-item questionnaire assessing pediatric peer relationships. Each item is rated on a scale from 1 (never) to 5 (almost always). A raw score is calculated based on the sum of item responses. The raw score is converted to a T-score ranging from 0-100, with a mean of 50 and a standard deviation of 10. Higher scores indicate stronger peer relationships.
Change in PROMIS Pediatric Item Bank v1.0 - Family Relationships - Short Form 8a | Baseline, Week 8
  This is an 8-item questionnaire assessing pediatric family relationships. Each item is rated on a scale from 1 (never) to 5 (always). A raw score is calculated based on the sum of item responses. The raw score is converted to a T-score ranging from 0-100, with a mean of 50 and a standard deviation of 10. Higher scores indicate stronger family relationships.
Change in PROMIS Pediatric Item Bank v1.0 - Sleep Disturbance - Short Form 8a | Baseline, Week 8
  This is an 8-item questionnaire assessing pediatric sleep disturbance. Each item is rated on a scale from 1 (never) to 5 (always). A raw score is calculated based on the sum of item responses. The raw score is converted to a T-score ranging from 0-100, with a mean of 50 and a standard deviation of 10. Higher scores indicate more prevalent sleep disturbance.
Change in School Engagement Scale Score | Baseline, Week 8
  23-item questionnaire assessing engagement in school. Each item is rated on a 6-point scale ranging from 1-5. The total score is the sum of responses and ranges from 23 to 115. Higher scores indicate greater school engagement.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Van Meter, PhD, Principal Investigator — NYU Langone Health; Erum Nadeem, PhD, Principal Investigator — Rutgers University
Locations (3):
- United States (3):
  - Rutgers University, New Brunswick, New Jersey
  - NYU Langone Health, Brooklyn, New York
  - Northwell Health School Mental Health Partnership sites, Glen Oaks, New York

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared with investigators whose proposed use of the data has been approved by the NIMH Data Archive. Data will be made available following article publication or as required by a condition of awards and agreements supporting the research. Data are available indefinitely through the NIMH Data Archive. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by the NIMH Data Archive will be shared to achieve aims in the approved proposal. Data are available indefinitely through the NIMH Data Archive.